CLINICAL TRIAL: NCT00197808
Title: Response of United Kingdom (UK) Infants to a Reduced Primary Schedule With Meningococcal C and Pneumococcal Conjugate Vaccines
Acronym: sched1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Public Health England (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: sched1
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2020-10-01 (Actual); Status verified 2018-08

CONDITIONS: Pneumococcal Infections; Meningococcal Infections
Keywords: Streptococcus pneumoniae; Neisseria meningitidis
MeSH Terms: conditions — Pneumococcal Infections; Meningococcal Infections

ARMS (6):
- Vaccine schedule 1 (Experimental): Menjugate vaccine at 2 and 3 months
  Interventions: Biological: menjugate
- Vaccine schedule 2 (Experimental): Menjugate vaccine at 2 and 4 months
  Interventions: Biological: Men C conjugate vaccine
- vaccine schedule3 (Experimental): Neissvacc at 2 and 3 months
  Interventions: Biological: Men C conjugate
- vaccine schedule 4 (Experimental): Neissvacc at 2 and 4 months
  Interventions: Biological: Men C Conjugate
- Vaccine schedule 5 (Experimental): Meningitec at 2 and 3 months
  Interventions: Biological: Men C conjugate
- Vaccine schedule 6 (Experimental): Meningitec at 2 and 4 months
  Interventions: Biological: Men C conjugate

INTERVENTIONS:
Biological: menjugate — men C conjugate vaccine
  Arms: Vaccine schedule 1
Biological: Men C conjugate vaccine — men C conjugate vaccine
  Arms: Vaccine schedule 2
Biological: Men C conjugate — men C conjugate vaccine
  Arms: vaccine schedule3
Biological: Men C Conjugate — men C conjugate vaccine
  Arms: vaccine schedule 4
Biological: Men C conjugate — men C conjugate vaccine
  Arms: Vaccine schedule 5
Biological: Men C conjugate — men C conjugate vaccine
  Arms: Vaccine schedule 6

SUMMARY:
The purpose of the study is to evaluate the immune responses of UK infants after one or two doses of pneumococcal conjugate vaccine or one or two doses of three different types of meningococcal conjugate vaccine given at either two and three or two and four months of age.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from parent or legal guardian of infant
* Age 7-11 weeks at first dose

Exclusion Criteria:

* Any contraindications to vaccination as specified in the UK Handbook "Immunisation Against Infectious Disease" (Ed 1996)
* < 7 weeks or > 11 weeks at first dose

Ages: 7 Weeks to 11 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 392 (Actual)
Dates: Start 2005-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Immunogenicity | 3 months after last sample
  SBA men C responses

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Coates, PhD, Study Chair — Public Health England
Locations (2):
- United Kingdom (2):
  - Hertfordshire Primary Care Trusts, Welwyn Garden City, Hertfordshire
  - Gloucestershire Primary Care Trusts, Gloucester

REFERENCES:
- [Result] Goldblatt D, Southern J, Ashton L, Richmond P, Burbidge P, Tasevska J, Crowley-Luke A, Andrews N, Morris R, Borrow R, Cartwright K, Miller E. Immunogenicity and boosting after a reduced number of doses of a pneumococcal conjugate vaccine in infants and toddlers. Pediatr Infect Dis J. 2006 Apr;25(4):312-9. doi: 10.1097/01.inf.0000207483.60267.e7. PMID 16567982
- [Derived] Goldblatt D, Southern J, Ashton L, Andrews N, Woodgate S, Burbidge P, Waight P, Miller E. Immunogenicity of a reduced schedule of pneumococcal conjugate vaccine in healthy infants and correlates of protection for serotype 6B in the United Kingdom. Pediatr Infect Dis J. 2010 May;29(5):401-5. doi: 10.1097/INF.0b013e3181c67f04. PMID 20010312
- See also: Published study results — https://www.ncbi.nlm.nih.gov/pubmed/16567982